CLINICAL TRIAL: NCT07161115
Title: A Phase II Study Evaluating the Efficacy and Safety of Neoadjuvant Therapy With MRI-Guided Involve-site Short-Course Radiotherapy Combined With Immunotherapy and Chemotherapy for Locally Advanced Rectal Cancer
Brief Title: Involve-site Radiotherapy Combined With Chemotherapy and Immunotherapy as Neoadjuvant Treatment for Locally Advanced Rectal Cancer
Acronym: REFIRT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Longhao Li (Other)
Responsible Party: Sponsor-Investigator, Longhao Li, M.D., First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1stChongqingMU-LLi
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Rectal Adenocarcinoma
Keywords: rectal cancers; radiotherapy; immunotherapy; Reducing the radiation field for radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Involve-site Short-Course Radiotherapy (Experimental)
  Interventions: Radiation: Reduced-field short-course radiotherapy; Drug: Immunotherapy combined with chemotherapy
- Standard long-course radiotherapy (Active Comparator)
  Interventions: Radiation: Standard long-course radiotherapy; Drug: Chemotherapy
- Standard short-course radiotherapy (Active Comparator)
  Interventions: Drug: Immunotherapy combined with chemotherapy; Radiation: Standard short-course radiotherapy

INTERVENTIONS:
Radiation: Reduced-field short-course radiotherapy — A dose of 25 Gy in 5 fractions was delivered as short-course radiotherapy, with one fraction per day, completing treatment within one week. The target volume was delineated using both CT and MRI. Compared to conventional radiotherapy fields, the irradiated volume was significantly reduced to include only the primary tumor and any metastatic lymph nodes as identified on MRI and CT.
  Arms: Involve-site Short-Course Radiotherapy
Drug: Immunotherapy combined with chemotherapy — After completion of radiotherapy, chemotherapy with the XELOX regimen (oxaliplatin 130 mg/m² on day 1 plus capecitabine 1500 mg/m² on days 1-14, every 3 weeks) was initiated in combination with sintilimab immunotherapy (200 mg every 3 weeks) for 4 cycles.
  Arms: Involve-site Short-Course Radiotherapy; Standard short-course radiotherapy
Radiation: Standard short-course radiotherapy — "Patients in the standard short-course radiotherapy group will receive 25 Gy in 5 fractions, once daily. Target volumes will be delineated according to the 2023 Guidelines for Target Volume Delineation and Planning of Rectal Cancer (National Cancer Center/National Cancer Quality Control Center), including the primary tumor, mesorectal region, and internal iliac and obturator lymph node drainage areas."
  Arms: Standard short-course radiotherapy
Radiation: Standard long-course radiotherapy — Patients in the standard long-course radiotherapy group will receive 50 Gy in 25 fractions, once daily, five days per week, with concurrent oral capecitabine chemotherapy. Target volumes will be delineated according to the 2023 Guidelines for Target Volume Delineation and Planning of Rectal Cancer (National Cancer Center/National Cancer Quality Control Center), including the primary tumor, mesorectal region, and internal iliac and obturator lymph node drainage areas.
  Arms: Standard long-course radiotherapy
Drug: Chemotherapy — Two weeks after the completion of radiotherapy, patients will receive four cycles of CAPOX chemotherapy.
  Arms: Standard long-course radiotherapy

SUMMARY:
Surgery is the primary treatment for rectal cancer. However, in patients with locally advanced disease, direct surgery often fails to achieve complete tumor resection. In such cases, neoadjuvant therapy is required to downstage the tumor before surgery. The current standard neoadjuvant approach consists of preoperative radiotherapy and then surgery. Although effective, standard radiotherapy uses large target volumes, which results in significant toxicities, increased surgical complications, and reduced patient compliance and quality of life. In addition, excessive radiation fields can compromise the intensity and timing of systemic therapy, potentially increasing the risk of distant metastasis. This may be one of the key reasons why current neoadjuvant radiotherapy mainly improves local control but has not translated into prolonged overall survival.

Emerging evidence suggests that combining immunotherapy with radiotherapy may further enhance treatment efficacy. However, large radiation fields may impair the effectiveness of immunotherapy. Therefore, reducing the radiotherapy target volume may not only decrease treatment-related toxicity but also augment the immunotherapy response.

This clinical study is designed to evaluate whether reducing the radiotherapy target volume, when combined with chemotherapy and immunotherapy prior to surgery, can decrease radiotherapy-related toxicities and reduce the risk of distant metastasis, without increasing the local recurrence rate, compared with the current standard radiotherapy fields. The ultimate goal is to improve the efficacy of neoadjuvant therapy in locally advanced rectal cancer while minimizing treatment toxicity, thereby providing new strategies and evidence for preoperative management.

DETAILED DESCRIPTION:
This study aims to provide stronger clinical evidence for involve-site short-course radiotherapy combined with immunotherapy as a neoadjuvant treatment strategy for locally advanced rectal cancer. The rationale for this trial is based on the limitations of standard radiotherapy, which uses large target volumes and results in significant toxicities, higher surgical complication rates, decreased patient compliance, reduced quality of life, and potentially compromised systemic therapy intensity. Reducing the radiation field is expected to lower treatment-related toxicity while preserving local tumor control and enhancing the efficacy of combined immunotherapy.

Study Objectives and Expected Outcomes The primary objective is to evaluate the safety and efficacy of involve-site short-course radiotherapy combined with chemotherapy and immunotherapy in patients with locally advanced rectal cancer, compared with conventional standard-field radiotherapy. The expected outcome is that the experimental regimen will demonstrate better safety, comparable or improved surgical resection and local control rates, and no higher incidence of distant metastasis relative to standard approaches.

Study Design and Methods This is a single-center, randomized, prospective, exploratory interventional trial. Due to the nature of the treatment, blinding is not feasible; thus, patients will be randomized in an open-label manner. Stratified randomization will be performed using block randomization with a block size of 6, and random sequences will be generated by the data management team.The study population will consist of 60 eligible patients who will be randomly assigned in equal numbers to three treatment groups (A, B, and C; 20 patients per group).

Group A (Control 1): Standard long-course radiotherapy (50 Gy in 25 fractions) combined with concurrent capecitabine chemotherapy, followed by four cycles of CAPOX chemotherapy and surgery, then four cycles of adjuvant CAPOX.

Group B (Control 2): Standard short-course radiotherapy (25 Gy in 5 fractions), followed two weeks later by four cycles of CAPOX chemotherapy plus sintilimab (anti-PD-1 immunotherapy), then surgery, followed by four cycles of adjuvant CAPOX.

Group C (Experimental): Involve-site short-course radiotherapy (25 Gy in 5 fractions), with the target volume limited to the primary tumor and involved lymph nodes as defined by MRI and CT imaging. One week after radiotherapy, patients will receive four cycles of CAPOX plus sintilimab, followed by surgery and then four cycles of adjuvant CAPOX.

Endpoints Primary Endpoint: Two-year local control rate (defined as the proportion of patients without pelvic recurrence or distant metastasis within 2 years after surgery).

Secondary Endpoints: Pathological complete response (pCR) rate, surgical resection rate, incidence of grade ≥3 radiation-induced proctitis, overall survival (OS), objective response rate (ORR), disease control rate (DCR), and incidence of severe postoperative complications (including anastomotic leakage, unplanned stoma, delayed wound healing beyond one month, severe infection, or thrombosis).

Patient Selection and Eligibility Eligible patients are those aged 18-75 years with histologically confirmed rectal adenocarcinoma, clinical stage T3-T4 and/or N+, and/or CRM-positive disease without lateral lymph node metastasis, and ECOG performance status of 0-1. Patients must not have received prior anticancer therapy and must provide signed informed consent.

Treatment and Follow-up Procedures Patients will undergo pre-treatment evaluation including physical examination, complete blood count, liver and renal function tests, tumor markers, electrocardiogram, pelvic MRI, and chest/abdominal contrast-enhanced CT. Follow-up evaluations will be performed every 3 months after surgery, and will continue until 24 months after the last patient undergoes surgery.

Data Collection and Outcome Assessment Tumor regression will be evaluated by MRI and pathological assessment according to Mandard tumor regression grading (TRG1-TRG5). Response will also be assessed by RECIST version 1.1 criteria.

Objective Response Rate (ORR): proportion of patients with CR or PR. Disease-Free Survival (DFS): time from surgery to recurrence, metastasis, or death.

Disease Control Rate (DCR): proportion of patients with CR, PR, or SD. Duration of Response (DOR): interval from initial response to progression or death.

Overall Survival (OS): time from randomization to death from any cause. Safety will be monitored and graded according to CTCAE version 5.0. The incidence, severity, and relationship of all adverse events (AEs), treatment-emergent AEs (TEAEs), serious AEs (SAEs), and immune-related AEs (irAEs) will be recorded. The number and proportion of patients requiring treatment modification or discontinuation due to AEs will be documented.

Statistical Analysis This exploratory trial will use a fixed sample size of 60 patients. Descriptive statistics will be used to summarize baseline characteristics. Continuous variables will be expressed as mean ± SD or median (range), while categorical variables will be summarized as frequency (percentage).

Study Timeline Planned enrollment period: 6 months. Planned follow-up: 24 months post-surgery. Total study duration: approximately 3 years. Study initiation: September 2025. Expected completion: August 2028.

Conclusion This trial is designed to evaluate whether involve-site short-course radiotherapy combined with chemotherapy and immunotherapy can achieve comparable local control while reducing toxicity and improving systemic outcomes in patients with locally advanced rectal cancer. The results are expected to provide new clinical evidence supporting optimized neoadjuvant strategies .

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agrees to participate and provides written informed consent
* Age 18 to 75 years, male or female
* Histologically confirmed rectal adenocarcinoma
* MRI confirms that the upper margin of the tumor is ≤12 cm from the anal verge
* ECOG performance status of 0-1
* Clinical stage T3-T4 or N+ and circumferential resection margin (CRM) positive by imaging evaluation; lateral lymph nodes negative
* Immunohistochemistry or genetic testing indicates pMMR or MSS status
* Adequate organ function and bone marrow reserve

Exclusion Criteria:

* Presence of distant metastasis
* Prior pelvic radiotherapy
* Chemotherapy or immunotherapy within the past 3 months
* Refusal to undergo radical surgery for rectal cancer
* Concurrent active malignancy other than rectal cancer
* Positive antinuclear antibody (ANA)
* History of autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, autoimmune hepatitis)
* Elevated troponin above the normal range
* Active tuberculosis
* Positive hepatitis B surface antigen (HBsAg) or detectable HBV DNA
* Positive for hepatitis C virus (HCV), syphilis, or HIV
* Severe comorbid conditions (e.g., serious infection, severe bone marrow suppression, psychiatric disorder) deemed unsuitable for participation by the investigator
* Pregnant or breastfeeding women
* Any other contraindications to radiotherapy, chemotherapy, or immunotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-19 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Two-year local control rate after rectal cancer surgery | At two years post-surgery
  Incidence of pelvic recurrence or distant metastasis within 2 years after surgery among the enrolled cohort

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) Rate | At the time of surgery
  Proportion of patients achieving pathological complete response (pCR) after neoadjuvant treatment.
Resection Rate | At the time of surgery
  Proportion of patients who undergo surgical resection after neoadjuvant therapy
Incidence of Grade ≥3 Radiation-induced Proctitis | From the start of radiotherapy until 2 years after surgery
  Number and proportion of patients experiencing grade 3 or higher radiation-induced proctitis, assessed according to CTCAE criteria.
Overall Survival (OS) | Up to 5 years after surgery
  Time from surgery to death from any cause.
Objective Response Rate (ORR) | From baseline until surgery
  Proportion of patients achieving complete response (CR) or partial response (PR), evaluated by RECIST 1.1 criteria.
Disease Control Rate (DCR) | From baseline until surgery
  Proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD), evaluated by RECIST 1.1 criteria.
Incidence of Severe Postoperative Complications | Within 30 days after surgery.
  Number and proportion of patients experiencing severe postoperative complications, including anastomotic leakage, unplanned stoma, wound healing delay >1 month, severe infection, or thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Longhao Li, M.D., Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared: De-identified participant data including demographics, treatment details (radiotherapy and chemotherapy), and efficacy and safety outcomes.
  Supporting documents: Study protocol, statistical analysis plan, and redacted informed consent forms.
  Start and end dates for data availability: Data available 6 months after primary results publication, for 5 years.
  Access criteria: Available to researchers with a scientifically sound proposal. Requests reviewed by the study steering committee; a data use agreement must be signed.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data available 6 months after primary results publication, for 5 years.
Access Criteria: Available to researchers with a scientifically sound proposal. Requests reviewed by the study steering committee; a data use agreement must be signed.